CLINICAL TRIAL: NCT04480710
Title: AMBITION: A Phase 2A, Multiple-Center, Single-Blind, Placebo-Controlled Study To Evaluate The Safety and Tolerability of CRV431 Dosed Once Daily in NASH Induced F2 and F3 Subjects
Brief Title: A Study of CRV431 Dosed Once Daily in NASH Induced F2 and F3 Subjects
Acronym: AMBITION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hepion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HEPA-CRV431-201
Record Dates: First submitted 2020-07-09; First posted 2020-07-21 (Actual); Results first posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-06

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; Fibrosis, Liver; NAFLD - Nonalcoholic Fatty Liver Disease
Keywords: Anti-fibrotic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — CRV-431

STUDY DESIGN:
Intervention Model Description: Randomized, multi-center, single-blind
Who Masked: Participant
Masking Description: placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CRV431 75mg (Experimental): CRV431, softgel capsule, 75mg, QD, 28 days, fasted conditions
  Interventions: Drug: CRV431 75mg
- Placebo, 75mg (Placebo Comparator): Placebo, softgel capsule, QD, 28 days, fasted conditions
  Interventions: Drug: Placebo (1 softgel)
- CRV431 225mg (Experimental): CRV431, softgel capsule, 225mg, QD, 28 days, fasted conditions
  Interventions: Drug: CRV431 225mg
- Placebo, 225mg (Placebo Comparator): CRV431, 3 softgel capsules, 225mg, QD, 28 days, fasted conditions
  Interventions: Drug: Placebo (3 softgels)

INTERVENTIONS:
Drug: CRV431 75mg — 1 x 75mg softgel capsule
  Arms: CRV431 75mg
Drug: Placebo (1 softgel) — 1 x placebo softgel capsule
  Arms: Placebo, 75mg
Drug: CRV431 225mg — 3 x 75mg softgel capsule
  Arms: CRV431 225mg
Drug: Placebo (3 softgels) — 3 x placebo softgel capsule
  Arms: Placebo, 225mg

SUMMARY:
This is a randomized, single-blind, placebo-controlled, once daily (QD) dose study of CRV431 in presumed NASH F2/F3 subjects.

DETAILED DESCRIPTION:
This is a randomized, single-blind, placebo-controlled, once daily (QD) dose study of CRV431 in presumed NASH F2/F3 subjects. Study will evaluate the safety and tolerability of a once daily 75mg dose and 225mg of CRV431 compared to placebo over 28 days of dosing. Pharmacokinetic parameters of CRV431 and its major metabolites and fraction unbound will also be evaluated. Non-invasive antifibrotic bio-markers will be collected and quantified from presumed NASH F2/F3 subjects dosed with 75mg CRV431 or placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female between 18 and 75 years of age (inclusive).
* Capable of giving written informed consent and able to effectively communicate with the investigator and study personnel.
* Presumed F2/F3 NASH to include: AST >20 IU/L, Pro-C3 >15.5 ng/mL, enhanced liver fibrosis (ELF) score >9.8, and FibroScan >8.5 kPa values.

Key Exclusion Criteria:

* Pregnant or breastfeeding or planning to become pregnant during the study period.
* Known allergy to CRV431, cyclosporine, or any of their inactive ingredients.
* Positive test for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCVAb) or human immunodeficiency virus antibodies (HIVAb).
* Well documented causes of chronic liver disease according to standard diagnostic procedures to include any history or presence of decompensated cirrhosis.
* Subjects with a platelet count <150,000/mL.
* Subjects with hemoglobin A1c(HbA1c) >9.5%.
* Weight loss of more than 5% within 3 months prior to randomization.
* Subjects with a blood pressure to include a systolic pressure >150 or a diastolic pressure >90.
* At Screening, an estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 mL (calculated by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] method) and/or a Kidney Disease Improving Global Outcomes (KDIGO) category of >G2.
* Subjects with a history of organ transplantation. Corneal transplantation will be allowed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Canizares, R.Ph., Study Director — Hepion Pharmaceuticals, Inc.
Locations (10):
- United States (9):
  - Conquest Clinical Research, Orange, California
  - Alliance Clinical Research, Poway, California
  - La Salud Research, Inc., Miami, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Covenant Research, LLC., Sarasota, Florida
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Aventiv Research Inc., Columbus, Ohio
  - Quality Research Inc., San Antonio, Texas
  - Pinnacle Research Group, San Antonio, Texas
- FDI Clinical Research, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo, 75mg | CRV431 75mg | Placebo, 225mg | CRV431 225mg
Started | 6 | 15 | 9 | 17
Completed | 6 | 12 | 8 | 17
Not Completed | 0 | 3 | 1 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRV431 75mg | Placebo, 75mg | CRV431 225mg | Placebo, 225mg | Total
Number analyzed (Participants) | 15 | 6 | 17 | 9 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (9.9) | 61.8 (8.7) | 54 (13.3) | 61.1 (13.8) | 58.0 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 10 | 2 | 23
  Male | 7 | 3 | 7 | 7 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 10 | 6 | 25
  Not Hispanic or Latino | 9 | 3 | 7 | 3 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 14 | 5 | 17 | 9 | 45
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
BMI [Mean (Standard Deviation); unit: kg/m^2] | 37.1 (8.5) | 36.1 (6.5) | 37.7 (6.4) | 39.2 (10.6) | 37.57 (7.82)
ALT [Mean (Standard Deviation); unit: IU/mL] | 62.5 (42.1) | 75.8 (36.8) | 39.3 (18.4) | 52.9 (35.6) | 51.46 (32.18)
AST [Mean (Standard Deviation); unit: IU/mL] | 51.9 (35.3) | 70.2 (40.1) | 33.1 (14.3) | 44.7 (36) | 43.83 (27.71)
Pro-C3 [Mean (Standard Deviation); unit: ng/mL] — Population: Missing baseline value
  ng/mL
    number analyzed (Participants) | 15 | 5 | 14 | 8 | 42
    (all) | 23.15 (6.88) | 23.19 (10.55) | 19.94 (9.07) | 18.56 (5.84) | 22.70 (12.44)
ELF Score [Mean (Standard Deviation); unit: units on a scale] — Calculated from three markers of fibrosis, hyaluronic acid, tissue inhibitor of matrix metalloproteinase-1 and aminoterminal propeptide of procollagen type III.
  Lower Risk: < 9.8 Mid Risk: 9.8 - 11.29 Higher Risk: >11.30
  The ELF Score is a unitless numerical value. *Harrison SA, Wong VW, Okanoue T, et al. Selonsertib for patients with bridging fibrosis or compensated cirrohsis due to NASH: Results from randomized phase III STELLAR trials. J Hepatol. 2020 Jul;73 (1) : 26-39.
  units on a scale | 10.3 (0.8) | 10.1 (0.4) | 9.8 (0.9) | 9.7 (1.0) | 10.0 (0.74)

OUTCOME MEASURES:

1. Primary Outcome: Number of Safety and Tolerability Events of CRV431 Versus Placebo.
Description: Number of adverse events, serious adverse events, and clinical laboratory abnormalities.
Time Frame: Time from informed consent to study day 42.
Population: Safety population.
Measure: Number; unit: Number of treatment emergent AE
Arm/Group | Placebo, 75mg | CRV431 75mg | Placebo, 225mg | CRV431 225mg
Number analyzed (Participants) | 6 | 15 | 9 | 17
Number of treatment emergent AE
  Number of Treatment Emergent Adverse Events | 4 | 8 | 3 | 21
  Relationship-unrelated | 4 | 6 | 2 | 13
  Relationship-possibly related | 0 | 0 | 1 | 1
  Relationship-probably related | 0 | 2 | 0 | 7
  Severity-Mild Grade 1 | 4 | 3 | 2 | 16
  Severity-Moderate Grade2 | 0 | 5 | 1 | 4
  Severity-Severe Grade 3 | 0 | 0 | 0 | 1
  Severity-Grade 4 | 0 | 0 | 0 | 0
  Number of Treatment Emergent Adverse Events leading to study withdrawl | 0 | 1 | 0 | 0

2. Primary Outcome: Tmax, of Once Daily (QD) 75mg and 225mg mg Doses of CRV431 is Presumed Non-alcoholic Steatohepatitis F2/F3 Fibrosis Subjects.
Description: The Tmax value is defined as time to reach maximum whole blood concentration. Each value is a median for the cohort along with the standard deviation presented in hours for Day 1 and Day 28.
Time Frame: Day 1 and Day 28
Measure: Median (Standard Deviation); unit: hours
Groups:
- 75 mg, Day 1; 75 mg, Day 28: 1 softgel capsule
- 225 mg, Day 1; 225 mg, Day 28: 3 softgel capsules
Arm/Group | 75 mg, Day 1 | 75 mg, Day 28 | 225 mg, Day 1 | 225 mg, Day 28
Number analyzed (Participants) | 15 | 15 | 17 | 17
hours | 4.41 (1.6) | 4 (2.05) | 2.59 (1.54) | 2 (0.73)

3. Primary Outcome: Cmax, of Once Daily (QD) 75mg and 22mg mg Doses of CRV431 is Presumed Non-alcoholic Steatohepatitis F2/F3 Fibrosis Subjects.
Description: The Cmax value is defined as the maximum whole blood concentration presented as ng/mL. Each value is a geometric mean for the cohort along with the standard deviation for Day 1 and Day 28.
Time Frame: Day 1 and Day 28
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | 75 mg, Day 1 | 225 mg, Day 1 | 75 mg, Day 28 | 225 mg, Day 28
Number analyzed (Participants) | 15 | 17 | 15 | 17
ng/mL | 347.24 (168.26) | 1147.31 (389.09) | 1218.88 (302.25) | 1876.9 (118.19)

4. Primary Outcome: AUC 0-last, of Once Daily (QD) 75mg and 225mg mg Doses of CRV431 in Presumed Non-alcoholic Steatohepatitis F2/F3 Fibrosis Subjects.
Description: The AUC 0-last value is defined as the area under the whole blood concentration time curve from time 0 to the time of the last measurable concentration. Each value is a geometric mean for the cohort along with the standard deviation for Day 1 and Day 28.
Time Frame: Timepoints for data collection include 0, 2.0 hours, 4.0 hours, 8 hours on both Day 1 and Day 28.
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 75 mg, Day 1 | 75 mg, Day 28 | 225 mg, Day 1 | 225 mg, Day 28
Number analyzed (Participants) | 15 | 15 | 17 | 17
h*ng/mL | 2251.32 (1054.20) | 8851.96 (2132.29) | 6348.85 (2819.58) | 13784.34 (4656.34)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of informed consent to day 42 of the study.
Arm/Group | CRV431 75mg | Placebo, 75mg | CRV431 225mg | Placebo, 225mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/6 | 0/17 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/6 | 0/17 | 0/9
Other Adverse Events (participants affected / at risk) | 5/15 | 3/6 | 10/17 | 3/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRV431 75mg (N=15) | Placebo, 75mg (N=6) | CRV431 225mg (N=17) | Placebo, 225mg (N=9)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Administration site condition
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SARS-CoV2 test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT04480710/Prot_SAP_001.pdf